CLINICAL TRIAL: NCT00940836
Title: Phase III Clinical Trial - Efficacy and Safety Assessment of a Compound Acetaminophen, Chlorpheniramine and Phenylephrine Combination in the Symptomatic Treatment of Common Cold and Flu-Like Syndrome in Adults
Brief Title: Efficacy and Safety Assessment of an Anti-Cold Preparation in the Symptomatic Treatment of Common Cold and Flu-Like Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Paulo Dornelles Picon, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05492
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2009-07

CONDITIONS: Common Cold; Flu-like Syndrome
Keywords: Anti-cold; Cold preparation; RCT
MeSH Terms: conditions — Common Cold | interventions — Acetaminophen; Chlorpheniramine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resfenol (Active Comparator): Patients in this arm will receive 15 capsules containing a combination described below. They are instructed to take one capsule at 7, 11, 15, 19 and 23h every day, starting after baseline evaluation. The duration of the treatment goes from 48 to 72 hours, depending on patient availability for the second evaluation.
  Patients also receive co interventional acetaminophen pills, that they are allowed to take in case of persisting pain or fever, up to 4 times a day.
  Interventions: Drug: Resfenol; Drug: Co interventional acetaminophen
- Placebo (Placebo Comparator): Patients in this arm will receive 15 capsules of placebo, that they are instructed to take in the same posology and in the same duration than the active comparator.
  Patients also receive co interventional acetaminophen pills, that they are allowed to take in case of persisting pain or fever, up to 4 times a day.
  Interventions: Drug: Placebo; Drug: Co interventional acetaminophen

INTERVENTIONS:
Drug: Resfenol — Each capsule of the active drug contains 400mg of acetaminophen, 4mg of chlorpheniramine and 4mg of phenylephrine. Patients will receive up to five capsules a day.
  Other Names: Anti-cold preparation; Acetaminophen; Chlorpheniramine; Phenylephrine
  Arms: Resfenol
Drug: Placebo — Patients in this group will receive placebo capsules up to five times a day, with the exact same taste and appearance as the active comparator.
  Arms: Placebo
Drug: Co interventional acetaminophen — All patients received, along with the assigned intervention, 12 acetaminophen 500mg pills, that they were instructed to take only in case of persisting PAIN or FEVER, up to 4 times a day.
  Other Names: Rescue medication; Acetaminophen; Paracetamol; Co intervention

SUMMARY:
The aim of this study is to assess the efficacy and safety of an anti-cold preparation compounded by acetaminophen, chlorpheniramine and phenylephrine for the treatment of cold and flu symptoms in healthy individuals in a randomized, double-blind, placebo-controlled clinical trial.

DETAILED DESCRIPTION:
Upper respiratory infections are rather frequent in the population, and their treatment consists, in most cases, in the use of symptomatic drugs. Acetaminophen is widely used as an analgesic and antipyretic, whereas chlorpheniramine is an antihistaminic and phenylephrine is a vasoconstrictor with decongestioning activity. The aim of this study is to assess the efficacy and safety of an anti-cold preparation, currently commercialized in Brazil by the name Resfenol, compounded by acetaminophen, chlorpheniramine and phenylephrine for the treatment of cold and flu symptoms in healthy individuals in a randomized, double-blind, placebo-controlled clinical trial.

Healthy volunteers are recruited through panels fixated at Hospital de Clínicas de Porto Alegre, in Brazil, and must answer a screening questionnaire at first contact. One hundred and forty six patients who met the inclusion criteria were included and, after baseline clinical and laboratory evaluation, were randomized to receive either the active intervention or placebo, 5 times a day, at 4 hour intervals, during 48 to 72 hours, depending on patient availability to show up for re-evaluation. Patients also received acetaminophen as a co intervention, to be taken only in case of persisting symptoms.

Patients answered, during treatment, several symptom questionnaires contained in a diary, and followup was performed at days 3 or 4 (clinical and laboratory evaluation) and 10 or 11 (clinical followup). Axillary temperature was assessed along with every dose with a thermometer provided by the study and registered in the diary.

Primary endpoint consists in the mean symptom scores, assessed through questionnaires in patient diary, baseline and followup. Secondary endpoints are global duration of symptoms, time of return to usual activities, use of co intervention for symptom relief, improval of fever and adverse effect evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 60 years old;
* Presenting with at least 6 and at max 72 hours of common cold symptoms (headache, muscle ache, rhinorrhea, nasal obstruction, sneezing, cough, sore or irritated throat, hoarseness, fever) or flu-like syndrome (high fever, muscle or articular ache, headache), with at least two symptoms rated by the patient as moderated to severe in an 0 to 4 scale;
* Proper anticonception, in the case of women in fertile age;
* Possibility to abstain from using any other drug for the treatment of the studied condition, except in emergencies, in wich case the responsible party must be immediately notified;
* Cooperation and understanding skills;
* Agreement to informed consent form.

Exclusion Criteria:

* Pregnant or lactating women;
* Hypersensitivity to any of the drug's components;
* Alcohol or substance abuse;
* Use of MAO inhibitor or barbituric;
* Diagnosis of any acute disease in current activity or uncontrolled chronic disease;
* Clinical evidence of immunosuppression;
* Influenza vaccine less than a week prior to inclusion;
* Need for antibiotic treatment for the respiratory infection, in the opinion of the investigator;
* Having participated in other clinical trial less than one year prior to inclusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Symptom improval assessed by questionnaires concerning headache, muscle ache, rhinorrhea, nasal obstruction, sneezes, cough, sore or irritated throat, hoarseness and fever, rated by patient himself in a scale from 0 to 4, being 0-absence and 4-severe. | Questionnaires were answered at baseline and 1st followup to the investigator and during treatment at every dose, 5 times a day, from day 1 to 3/4, through patient's diary.

SECONDARY OUTCOMES:
Global duration of symptoms, assessed by the investigator through direct questioning at followup visits. | Day 3/4 and, if no relief yet, day 10/11.
Time of return to usual activities, such as work or gym, assessed by the investigator through direct questioning at followup visits. | Day 3/4 and, if no relief yet, day 10/11.
Use of co intervention for symptom relief during treatment, registered by the volunteer in patient diary, with day and hour of ingestion. | Assessed during treatment (day 1 to 3/4) by patient diary and questioned by investigator at 1st followup visit.
Improval of fever by reduction of axillary temperature to less than 38,1°C. | Assessed by investigator at baseline and 1st followup visit and by patient (with termometer provided by the study) along with every dose, 5 times a day, from day 1 to 3/4, registered in patient diary.
Adverse effect appearance during and until 7 days after treatment, assessed through patient's report in the diary or followup visit, through physical evaluation at followup and by laboratory exams. | Days 1 to 3/4 through patient diary, and followup at days 3/4 an 10/11.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil